CLINICAL TRIAL: NCT06134284
Title: Prospective, Multicenter, Single-arm Clinical Study of Orelabrutinib Plus Rituximab for Second-line Treatment of Relapsed/Refractory Marginal Zone Lymphoma
Brief Title: Clinical Study of OR for Second-line Treatment of Refractory MZL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lixia Sheng (Other)
Responsible Party: Sponsor-Investigator, Lixia Sheng, hematology department, Ningbo No. 1 Hospital
Organization: Ningbo No. 1 Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ningbo102
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: OR Regimen for Relapsed/Refractory Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OR regimen (Experimental): The specific medication regimen for the OR regimen is as follows: Orelabrutinib 150mg orally once daily; Rituximab 375mg/m² intravenous infusion, administered every 21 days.
  Interventions: Drug: Orelabrutinib combined with rituximab

INTERVENTIONS:
Drug: Orelabrutinib combined with rituximab — This is a single-arm trial. Patients with relapsed/refractory marginal zone lymphoma will be treated with the OR regimen. The treatment plan is as follows: Orelabrutinib 150mg oral administration once a day, Day 1-21; Rituximab 375mg/m² intravenous infusion, Day 1. Each cycle is 21 days. PET-CT evaluation will be conducted after 4 cycles. If a partial response (PR) or better is achieved, the patient will receive further treatment with the OR regimen for an additional 4 cycles before transitioning to single-agent maintenance therapy with either rituximab or obinutuzumab. If a PR or better is not achieved after 4 cycles, the patient will discontinue from the trial.

SUMMARY:
The goal of this clinical trial is to test the overall response rate of Orelabrutinib combined with rituximab (OR regimen) for second-line treatment of relapsed/refractory marginal zone lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years, 80, Sex gender no limitied;
2. histological confirmation of MZL, For splenic marginal zone lymphoma (SMZL) where histological specimens of the spleen were not available, Requirements to meet the minimum diagnostic criteria for SMZL, And exclude any other type of small B cell lymphoma, That is, requiring a definite diagnosis of MZL;
3. at least one two-dimensional measurable lymph node lesion (CT scan or MR / display maximum diameter> 1.5cm), Or at least one two-dimensional measurable extranodal lesion (CT scan or MRI showing maximum diameter> 1.0cm);
4. the investigator required systemic treatment for marginal zone lymphoma;
5. at least 1 previous course of systemic lymphoma treatment (including previous immunotherapy or chemoimmunotherapy), 3 without efficacy above PR after imaging evaluation, Or disease progression after effective treatment;
6. ECOG, physical strength score 0-2;
7. primary organ function meets the following criteria 7 days prior to treatment:

   1. blood routine: absolute neutrophil ≥1.5x10^9 / L, Platelet≥ 75x10^9 / L, Hemoglobin≥75g / L; If the concomitant bone marrow invasion, Absolute neutrophil value ≥1.0x10^9 / L, Platelet≥50x10^9 / L, Hemoglobin≥ 50g / L;
   2. Blood Chemistry: total bilirubin ≤1.5 times ULN, AST or ALT ≤2 times ULN; If the liver is infiltrated with a lymphoma, Then, ALT and AST ≤5 times ULN, Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥45 ml/min (Cockcroft-Gault formula); Serum amylase ≤ULN;
   3. coagulation function: International normalized ratio (INR) ≤1.5 times ULN, Activated partial thromboplastin time (APTT)≤ 1.5 times ULN.
   4. cardiac color ultrasound: left ventricular ejection fraction 50%;
8. expected survival time of 3 months;
9. for men who did not undergo sterilization: agree to use the barrier contraceptive method during treatment and for at least 3 months after the last administration of obutinib or rituximab or on the older) as required in the guidelines established by the institution. In addition, male patients must agree to request their spouses to use other methods of contraception (e. g., oral contraceptives, intrauterine devices, barrier contraception, or spermicide).
10. For women who did not undergo sterilization: at least 28 days prior to consent to start study medication, during treatment, or after last administration of obutinib or rituximab, such as oral contraceptives, intrauterine devices or barrier contraception;
11. voluntarily signed written informed consent before test screening.

Exclusion Criteria:

1. The patient had been previously treated with obutinib in combination with rituximab, Efficacy was assessed as being refractory, Infraciness was defined as no remission (PR or CR) after start of treatment 4
2. history of severe allergy or allergic reaction to monoclonal antibody therapy
3. known to be allergic to any study drug
4. current or previous other malignancy, Unless curative treatment with no evidence of recurrence and metastasis in nearly 5 years;
5. lymphoma involvement of the central nervous system;
6. uncontrolled or important cardiovascular disease, Includes:

   1. occurrence of New York Cardiology Association (NYHA) grade II or above congestive heart failure, unstable angina, myocardial infarction within 6 months prior to the first administration of study drug, Or the presence of significant arrhythmias requiring treatment at screening (e. g., persistent rapid AF, persistent ventricular tachycardia, ventricular fibrillation, tip torsion, history of second-degree II AV (AV) block, or history of third-degree AV block), Left ventricular ejection fraction (LVEF) <50%;
   2. primary cardiomyopathy (e. g. dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, irregular cardiomyopathy);
   3. history of clinically significant QTc interval extension, Or subjects with coronary heart disease with QTc interval female> 470ms and male> 450ms;
   4. symptomatic or requiring medication;
   5. difficult-to-control hypertension (on the basis of improved lifestyle, With an adequate amount of 2 or more antihypertensive drugs (including diuretics) for more than 1 month, Or take 4 or more antihypertensive drugs to effectively control blood pressure).
7. Active bleeding within the 2 months prior to screening, Or are taking anticoagulant drugs, Or if the investigator considers a definite bleeding tendency;
8. urine protein 2 +, And 24-hour urinary protein quantification of 2g / 24 hours;
9. a history of deep vein thrombosis or pulmonary embolism;
10. clinically obvious gastrointestinal abnormalities, May affect drug intake, transport, or absorption (e. g. inability to swallow, chronic diarrhea, intestinal obstruction, etc.), Or subjects with total gastrectomy;
11. history of organ transplantation or allogeneic bone marrow transplantation;
12. major surgery within 6 weeks or minor surgery within 2 weeks before screening. Major surgery is using general anesthesia, but diagnostic endoscopy is not considered a major surgical procedure. The insertion of a vascular access device will be exempted from this exclusion criteria;
13. active infection or uncontrolled HBV (HBV DNA titer of 10 ^ 3 copies / ml), HCVAb positive, HI V/A IDS (Acquired Immune Deficiency Syndrome) or other serious infectious diseases;
14. subjects with current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc.;
15. Previous treatment with BTK, BCR, pathway inhibitors (such as PI3K, Syk), and BCL-2 kinase inhibitors;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 8 months
  Proportion of CR and PR subjects will be assessed at 8 courses

SECONDARY OUTCOMES:
Progress free survival time | up to36 months
  To measure the duration of response over a follow-up period of 36 months
Overall survival | up to36 months
  OS will be assessed from the first receptor given to death or last follow-up.
Adverse events profile | Measured from start of treatment until 21 days after last dose
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Chen, Principal Investigator — First Affiliated Hospital of Ningbo University
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Zhejiang University, Ningbo First Hospital, Hangzhou, Zhejiang
  - 86-574-87085596, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No